CLINICAL TRIAL: NCT04374786
Title: Effects of a Mobile App on Health and Well-being During COVID-19 Pandemic in House Staff at Banner University Medical Center Phoenix
Brief Title: Effects of Mobile App in House Staff Health and Well-being During COVID-19 Pandemic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss to follow up. No longer enrolling.
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Kelley Saunders, Clinical Assistant Professor, Principal Investigator, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2003524869 [Sub-study]
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Perceived Stress; Anxiety; Sleep Disturbance; Burnout; PTSD
Keywords: COVID-19; mindfulness meditation
MeSH Terms: conditions — Anxiety Disorders; Parasomnias; Burnout, Psychological; Stress Disorders, Post-Traumatic; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Will receive a 30-day are trial of the mobile meditation app "Calm" on study day 0
  Interventions: Device: Calm Meditation App

INTERVENTIONS:
Device: Calm Meditation App — Meditation is a self-management strategy that can be utilized by anyone to assist with the management of stress. Meditation mobile applications, such as the "Calm" app, can be used to help manage stress, especially during this uncertain time.

SUMMARY:
Due to the COVID-19 global health pandemic, many people are likely experiencing increased stress. The well-being of physicians in training may be significantly impacted by this pandemic. Meditation is a self-management strategy that can be utilized by anyone to assist with the management of stress. Meditation mobile applications, such as the "Calm" app, can be used to help manage stress, especially during this uncertain time. The investigators propose a prospective evaluation of perceived stress, anxiety, burnout and sleep disturbance in the house staff at Banner University Medical Center Phoenix, with the use of the mobile meditation app, "Calm." The investigatros additionally want to evaluate the feasibility of using the mobile app, including looking at adherence to use of the app and physician satisfaction with use of the app.

DETAILED DESCRIPTION:
The COVID-19 global pandemic is significantly impacting healthcare providers and presumably affecting their stress level as they deal with this time of uncertainty. The COVID-19 public health crisis requires the full resources and attention of healthcare systems. This has led to several healthcare changes that affect physicians in training, including changes to rotations and schedules, risks of infection exposure to themselves or their families, and the unknown impacts this may have on their residency and fellowship experiences.

These changes are likely impacting their stress, health, and well-being. Physician burnout is major concern for the medical community and likely to be further impacted by the current pandemic. Evidence-based interventions for stress include cognitive behavior therapy, although this can be time consuming, requires the need for specialized providers, and is not feasible for everyone during this COVID-19 pandemic. Pharmacotherapy can be used, including antidepressants and anxiolytics, however they have inherent limitations such as side effects, tolerance, and interactions that limit their use. Consumer based mobile applications (apps) may help individuals with self-management strategies for stress. Mindfulness meditation is one type of self-management strategy and is the practice of moment-to-moment awareness in which the person purposefully focuses on the present without judgement.

"Calm" is a mobile app that offers a range of meditation lessons, sleep stories (bed-time stories for grown-ups), sleep music, and nature sounds with modules that vary in length, instruction, and content. Few studies on the use of "Calm" exist and include a randomized controlled trial evaluating its affect to decrease stress among college students and a descriptive study evaluating cancer patient's perceptions of the app. There is evidence to support the use of similar apps in resident physicians. A pilot study assessing the effects of a meditation app on resident wellness suggested both the feasibility and efficacy of such an intervention. During these unprecedented times of the COVID-19 pandemic, mobile apps such as Calm may be potentially beneficial to help with stress in house staff physicians, although this requires further investigation.

ELIGIBILITY:
Inclusion Criteria:

* All resident and fellow physicians at Banner University Medical Center Phoenix, 1111 E. McDowell Rd, Phoenix, AZ 85006.

Exclusion Criteria:

* Non-resident and fellow physicians at Banner University Medical Center Phoenix, 1111 E. McDowell Rd, Phoenix, AZ 85006.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Completed study Day 0
  Validated perceived stress scale survey, 10 questions in length rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Individual scores can range from 0 to 40 with higher scores indicating higher perceived stress.
Perceived Stress Scale | Completed study Day 14
  Validated perceived stress scale survey, 10 questions in length rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Individual scores can range from 0 to 40 with higher scores indicating higher perceived stress.
Perceived Stress Scale | Completed study Day 30
  Validated perceived stress scale survey, 10 questions in length rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Individual scores can range from 0 to 40 with higher scores indicating higher perceived stress.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Completed study Day 0, 14, and study Day 30
  Validated anxiety and depression scale survey, 14 questions in length rated on a 4-point Likert scale. Possible scores range from 0 to 21 for anxiety and 0 to 21 for depression with higher scores indicating probable presence of the mood disorder.
PROMIS Sleep Disturbance Short Form Survey | Completed study Day 0, 14, and study Day 30
  Patient Reported Outcomes Measurement Information System (PROMIS) is a validated sleep disturbance short form survey, 8 questions in length rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (very much). Possible scores range from 0 to 21 for anxiety and 0 to 21 for depression with higher scores indicating greater severity of sleep disturbance.
Impact of Event Scale-6 | Completed study Day 0, 14, and study Day 30
  The Impact of Event Scale-6 is a validated post traumatic event survey, 6 questions in length rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (extremely). The score ranges from a minimum of 6 to a maximum of 30 with higher scores indicating higher traumatic stress.
Maslach Burnout Inventory | Completed study Day 0, 14, and study Day 30
  The Maslach Burnout Inventory is a validated burnout survey, 22 questions in length with 3 sub scales including emotional exhaustion, depersonalization, and personal accomplishment. Each question is rated on a 7 point Likert scale ranging from 0 (never) to 6 (every day). The score for each sub scales range from minimum 0 to maximum 18. High scores of emotional exhaustion and depersonalization sub scales and a lower score of personal accomplishment indicates a higher level of burnout.
Adherence | From Day 0 to Day 30
  Usage data from mobile app, minutes per day used
Coronavirus Questionnaire | Completed study Day 0 and study Day 30
  Investigator developed questionnaire about perceptions on coronavirus completed on Day 0 and Day 30, 10 questions in length and measured with 5-point Likert scale. 1= very low, 2=low, 3=moderate, 4=high, 5= very high.
Participant Satisfaction | Completed study Day 30
  Investigator developed satisfaction questionnaire completed on Day 30, 13 questions in length.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Foley, MD, Study Chair — Chair - BUMCP
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huberty J, Green J, Glissmann C, Larkey L, Puzia M, Lee C. Efficacy of the Mindfulness Meditation Mobile App "Calm" to Reduce Stress Among College Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 25;7(6):e14273. doi: 10.2196/14273. PMID 31237569
- [Result] Huberty J, Vranceanu AM, Carney C, Breus M, Gordon M, Puzia ME. Characteristics and Usage Patterns Among 12,151 Paid Subscribers of the Calm Meditation App: Cross-Sectional Survey. JMIR Mhealth Uhealth. 2019 Nov 3;7(11):e15648. doi: 10.2196/15648. PMID 31682582
- [Result] Huberty J, Puzia M, Eckert R, Larkey L. Cancer Patients' and Survivors' Perceptions of the Calm App: Cross-Sectional Descriptive Study. JMIR Cancer. 2020 Jan 25;6(1):e16926. doi: 10.2196/16926. PMID 32039812
- [Result] Wen L, Sweeney TE, Welton L, Trockel M, Katznelson L. Encouraging Mindfulness in Medical House Staff via Smartphone App: A Pilot Study. Acad Psychiatry. 2017 Oct;41(5):646-650. doi: 10.1007/s40596-017-0768-3. Epub 2017 Aug 9. PMID 28795335